CLINICAL TRIAL: NCT02741323
Title: Impact of CCR5 Blockade in HIV+ Kidney Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HIVTR-CCR5; 20730 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: HIV Infections; Kidney Diseases
Keywords: HIV-infected with end-stage kidney disease
MeSH Terms: conditions — HIV Infections; Kidney Diseases | interventions — Maraviroc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Maraviroc (MVC) (Experimental): Participants will receive MVC at the time of admission for transplantation and prior to transplant. Participants will receive MVC throughout their participation in the study, which will be 1 to 3 years depending on when they enroll.
  Interventions: Drug: Maraviroc
- Arm 2: Placebo (Placebo Comparator): Participants will receive placebo at the time of admission for transplantation and prior to transplant. Participants will receive placebo throughout their participation in the study, which will be 1 to 3 years depending on when they enroll.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Maraviroc — Initial dose of 300 mg twice daily (150mg twice daily if co-prescribed with a potent CYP3A inhibitor or 600mg twice daily if co-prescribed with a potent CYP3A inducer). Will be modified if GFR < 30, if co-prescribed with a potent CYP3A inhibitor or inducer, or if the calcineurin inhibitor used for maintenance immunosuppression is changed to cyclosporine (which is only allowed for tacrolimus toxicity).
  Once GFR is greater than or equal to 30, the dose should be returned to the non-renal dosage. If GFR is consistently fluctuating (especially immediately post-transplant), the site investigator may choose when to resume normal dosing of study product based on clinical assessment of stability.
  Other Names: MVC
  Arms: Arm 1: Maraviroc (MVC)
Drug: Placebo — Initial dose of 300 mg twice daily (150mg twice daily if co-prescribed with a potent CYP3A inhibitor or 600mg twice daily if co-prescribed with a potent CYP3A inducer). Will be modified if GFR < 30, if co-prescribed with a potent CYP3A inhibitor or inducer, or if the calcineurin inhibitor used for maintenance immunosuppression is changed to cyclosporine (which is only allowed for tacrolimus toxicity).
  Once GFR is greater than or equal to 30, the dose should be returned to the non-renal dosage. If GFR is consistently fluctuating (especially immediately post-transplant), the site investigator may choose when to resume normal dosing of study product based on clinical assessment of stability.
  Arms: Arm 2: Placebo

SUMMARY:
Maraviroc (MVC) is a type of HIV medicine called a CCR5 inhibitor. This study will evaluate the safety and tolerability of MVC in HIV-infected adults receiving a kidney transplant.

DETAILED DESCRIPTION:
MVC is a CCR5 inhibitor that may have a positive role in modulating the immune response following transplantation. The purpose of this study is to evaluate the safety and tolerability of MVC in HIV-infected adults in need of a kidney transplant. The study will also evaluate whether using both immunosuppressant drugs and MVC will improve kidney function after a kidney transplant.

This study will enroll HIV-infected adults on combination antiretroviral therapy (cART) who need a kidney transplant. At the time of their kidney transplant, study participants will be randomly assigned to receive either MVC or placebo as an addition to their cART regimen. (MVC or placebo will be provided by the study. However, the HIV medicines in their cART regimens will not be provided by the study.) Participants will receive MVC or placebo throughout their participation in the study, which will be 1 to 3 years depending on when they enroll in the study.

Study visits will occur at enrollment (Day 0) and post-transplant Weeks 1, 2, 4, 8, 13, 26, 39, 52, 78, 104, 130, and 156. Study visits may include a physical examination, blood collection, lymph node collection, urine sample collection, and a kidney biopsy. During the study, participants will also be monitored closely for evidence of drug toxicities, HIV treatment failure and rejection.

ELIGIBILITY:
Inclusion Criteria:

* Participant is able to understand and provide informed consent.
* Documented HIV infection (by any licensed enzyme-linked immunosorbent assay [ELISA] and confirmation by Western Blot, positive HIV antibody (ab) indirect fluorescent antibody (IFA), or documented history of detectable HIV-1 RNA).
* Participant is 18 years of age or older.
* CD4+ T-cell count greater than or equal to 200/µL at any time in the 26 weeks prior to enrollment.
* Most recent HIV-1 RNA less than 50 copies RNA/mL. Eligibility at the time of enrollment will be determined based on the most recent HIV-1 RNA, not more than 26 weeks prior to enrollment. Subjects who require a switch in combination antiretroviral therapy (cART) regimen to become study eligible must also have an eligible HIV-1 RNA result post change in cART.
* Participant meets standard listing criteria for placement on transplant waiting list.
* For participants with an HIV+ deceased donor:

  * No active opportunistic infections.
  * Concurrence by the study team that based on medical history and ART, viral suppression can be achieved in the recipient post-transplant.
  * Must be enrolled in an Institutional Review Board (IRB) approved research protocol that fulfills the requirements of the DHHA Hope Act Policy (see the protocol for more information).
  * HIV+ deceased donor must have no evidence of invasive opportunistic complications of HIV infection, and must have a pre-implant biopsy.
* Antiretroviral (ARV) Use: Participant is on a stable cART regimen for at least 3 months prior to enrollment (unless changes are made due to toxicity, drug interactions, convenience or to an eligible non-protease inhibitor-based regimen). Switch should not be due to virologic failure. A regimen consisting of 2 NTRTIs and an integrase inhibitor is preferred due to minimal drug interaction but any non-protease inhibitor regimen may be used.

  * If on a protease inhibitor based regimen, participant must be switched to a non-protease inhibitor-based regimen based on lack of any prior drug resistance or antiretroviral-treatment failure, and be willing to remain on indefinitely unless a change is medically necessary. Participants who need to be switched must have been on a stable cART regimen for at least 3 months prior, and must have an eligible HIV-1 RNA result post change in cART.
  * If already on a stable non-protease inhibitor-based regimen, participant is willing to remain on this regimen indefinitely unless a change in regimen is medically indicated.
  * If untreated, must initiate and be willing to remain on indefinitely a non-protease inhibitor-based antiretroviral regimen unless a change is medically necessary.
* No known allergy or intolerance to components of maraviroc (MVC) or its formulation.
* No known contraindication to MVC.
* Female participants of child-bearing potential must have a negative serum beta-human chorionic gonadotropin (HCG) pregnancy test within 30 days of randomization.

Exclusion Criteria:

* Participant is currently on MVC.
* Participant needs multi-organ transplant.
* Participant has a live donor who is HIV+.
* Participant is unable to switch to a non-protease inhibitor-based cART regimen.
* Participant has received immunosuppressant medication in the 6 months prior to enrollment. Note: Low dose maintenance steroids (less than or equal to 10 mg per day of prednisone, or equivalent strength steroid) will not be considered immunosuppression.
* Opportunistic Complication History: Any history of progressive multifocal leukoencephalopathy (PML), chronic intestinal cryptosporidiosis of greater than 1 month duration, or primary central nervous system (CNS) lymphoma. Note: History of pulmonary coccidioidomycosis will be treated per local site policy regarding this infection in HIV negative transplant candidates, generally requiring a 5-year disease-free interval.
* Participant has a history of any neoplasm except for the following: resolved kaposi's sarcoma, in situ anogenital carcinoma, adequately treated basal or squamous cell carcinoma of the skin, solid tumors (except primary CNS lymphoma) treated with curative therapy and disease free for more than 5 years. History of renal cell carcinoma requires disease-free state for 2 years. History of leukemia and disease-free duration will be per site policy.
* Substance use that in the opinion of the investigator would interfere with compliance with the study requirements.
* Participant is pregnant or breastfeeding. Note: Participants who become pregnant post-transplant will continue to be followed in the study and will be managed per local site practice. Women that become pregnant should not breastfeed.
* Participant has used interleukin-2 (IL-2) or granulocyte-macrophage colony-stimulating factor (GM-CSF) in the prior six months.
* Participant has received interferon-alpha therapy in the prior 12 weeks.
* Use of investigational drugs within 4 weeks of enrollment.
* Past or current medical problems or findings from medical history, physical examination, or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements, or that may impact the quality or interpretation of the data obtained from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stock, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (10):
- United States (10):
  - UAB HIVTR-CCR5 Non-Network CRS, Birmingham, Alabama
  - UCLA HIVTR-CCR5 Non-Network CRS, Los Angeles, California
  - UCSF HIVTR-CCR5 Non-network CRS, San Francisco, California
  - Georgetown HIVTR-CCR5 Non-Network CRS, Washington D.C., District of Columbia
  - Emory HIVTR-CCR5 Non-Network CRS, Atlanta, Georgia
  - Northwestern HIVTR-CCR5 Non-Network CRS, Chicago, Illinois
  - Univ. of Maryland HIVTR-CCR5 Non-Network CRS, Baltimore, Maryland
  - JHU HIVTR-CCR5 Non-Network CRS, Baltimore, Maryland
  - Mt. Sinai Med. Ctr. HIVTR-CCR5 Non-Network CRS, New York, New York
  - Univ. of Penn HIVTR-CCR5 Non-network CRS, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Maraviroc (MVC): Participants who were assigned to and received Maraviroc in the study.
- Arm 2: Placebo: Participants who were assigned to and received Placebo in the study.
Period: Overall Study
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Started | 49 | 48
Completed (Provided at least 1-year survival data, completing the requirement for at least 1-3 years of follow-up in the study) | 43 | 40
Not Completed | 6 | 8

BASELINE CHARACTERISTICS:
Population: The analysis population includes all subjects who were randomized, received at least 1 dose of Maraviroc or Placebo, and underwent kidney transplant.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 42 | 84
  >=65 years | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (10.8) | 53.1 (10.3) | 52.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 42 | 43 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 44 | 41 | 85
  Unknown or Not Reported | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 5 | 8 | 13
  Race: Black or African American | 39 | 36 | 75
  Race: Asian | 2 | 1 | 3
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Race: Unknown/ Not Reported | 2 | 1 | 3
  Race: Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 49 | 48 | 97

OUTCOME MEASURES:

1. Primary Outcome: Mean Glomerular Filtration Rate by Iohexol Clearance at Week 52
Description: The primary efficacy endpoint is the 52-week GFR as measured by iohexol clearance
Time Frame: Measured at Week 52 Post-transplant
Population: Included Full Analysis Population participants with available 52-week GFR level
Measure: Mean (95% Confidence Interval); unit: mL/min/1.73 m²
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 18 | 13
mL/min/1.73 m² | 37.0 [30.1 to 43.9] | 40.1 [26.9 to 53.3]

2. Primary Outcome: Cumulative Incidence of Graft Loss, Toxicities ≥ Grade 3 Per the DAIDS Toxicity Table and/or Permanent Treatment Discontinuation
Description: The primary safety endpoint will be the incidence of graft loss and toxicities ≥ Grade 3 and/or permanent treatment discontinuation within the first 52 weeks post-transplant
Time Frame: Measured through Week 52 Post-transplant
Measure: Number (95% Confidence Interval); unit: Proportion (KM estimate for incidence)
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 49 | 48
Proportion (KM estimate for incidence) | 0.84 [0.72 to 0.93] | 0.85 [0.74 to 0.94]

3. Secondary Outcome: Mean CD45 Gene Expression Count (PTPRC)
Description: Based on the formalin-fixed paraffin-embedded (FFPE) kidney biopsy sample. CD45 RNA In Situ Hybridization was performed, and the CD45 gene expression count is calculated by counting the "spots" (the RNA signal) in QuPath and then dividing the number of spots by biopsy tissue area in mm².
Time Frame: Measured at Week 26 Post-transplant
Population: Full Analysis Population
Measure: Median (Inter-Quartile Range); unit: spots/mm²
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 15 | 10
spots/mm² | 49.4 [12.3 to 129.0] | 50.9 [16.2 to 518.0]

4. Secondary Outcome: Mean CD45 Quantitative Immunohistochemistry (IHC)
Description: Mean CD45 quantitative immunohistochemistry (IHC) based on FFPE sample
Time Frame: Measured at Week 26 Post-transplant
Population: Full Analysis Population
Measure: Median (Inter-Quartile Range); unit: cells/mm²
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 20 | 15
cells/mm² | 144.7 [84.5 to 294.0] | 77.5 [15.0 to 285.9]

5. Secondary Outcome: Tissue Common Rejection Module (tCRM) Score Using the 11-gene tCRM Module on FFPE Biopsy Shaves
Description: Tissue Common Rejection Module (tCRM) score using the 11-gene tCRM module on FFPE biopsy shaves at 26 weeks. The score measures the average (geometric mean) gene expression level of CRM genes (BASP1, CD6, CXCL10, CXCL9, INPP5D, ISG20, LCK, NKG7, PSMB9, RUNX3, TAP1) in kidney tissue. Possible range (min-max) for the tCRM score is 0.01 - 15.0, with higher values representing worse outcomes.
Time Frame: Measured at Week 26 Post-transplant
Population: Full Analysis Population - subset of participants with available data at 26 weeks.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 23 | 21
score on a scale | 1.83 [1.09 to 3.36] | 1.67 [1.14 to 2.16]

6. Secondary Outcome: Urine Common Rejection Module (uCRM) Score Using the 11-gene uCRM Module on Urine Cell Pellets
Description: Urine Common Rejection Module (uCRM) score using the 11-gene uCRM module on urine cell pellets at week 26. The score measures the average (geometric mean) gene expression level of CRM genes (BASP1, CD6, CXCL10, CXCL9, INPP5D, ISG20, LCK, NKG7, PSMB9, RUNX3, TAP1) in urine sediment. Possible range (min-max) for the uCRM score is 0.01 - 15.0, with higher values representing worse outcomes.
Time Frame: Measured at Week 26 Post-transplant
Population: Full Analysis Population - subset of participants with available data at Week 26
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 24 | 21
score on a scale | 0.48 [0.23 to 1.08] | 0.42 [0.20 to 0.87]

7. Secondary Outcome: Urine Common Rejection Module (uCRM) Score Using the 11-gene uCRM Module on Urine Cell Pellets
Description: Urine Common Rejection Module (uCRM) score using the 11-gene uCRM module on urine cell pellets at week 52. The score measures the average (geometric mean) gene expression level of CRM genes (BASP1, CD6, CXCL10, CXCL9, INPP5D, ISG20, LCK, NKG7, PSMB9, RUNX3, TAP1) in urine sediment. Possible range (min-max) for the uCRM score is 0.01 - 15.0, with higher values representing worse outcomes.
Time Frame: Measured at Week 52 Post-transplant
Population: Full Analysis Population - subset of participants with available data at Week 52
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 21 | 17
score on a scale | 0.40 [0.12 to 0.85] | 0.25 [0.16 to 0.64]

8. Secondary Outcome: Proportion of Participants With Estimated Glomerular Filtration Rate (eGFR) Less Than 60 mL/Min/1.73 m² at Week 52
Description: Measured by Chronic Kidney Disease Epidemiology collaboration equation (CKD-EPI) Creatinine equation
Time Frame: Measured at Week 52 Post-transplant
Population: Full Analysis Population participants with available data at Week 52.
Measure: Number (95% Confidence Interval); unit: Proportion
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 44 | 37
Proportion | 0.45 [0.33 to 0.63] | 0.73 [0.60 to 0.89]

9. Secondary Outcome: Proportion of Participants With Defined CKD Stage 4 or 5 at Year 1
Description: Proportion of participants with defined CKD stage 4 or 5 at week 52 post-transplant. CKD Stage 4 or 5 is defined as a glomerular filtration rate (GFR) of <30 mL/min.
Time Frame: Year 1 time point
Population: Participants in the Full Analysis population with available data at Year 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 44 | 37
Proportion of participants | 0.07 [0.02 to 0.20] | 0.14 [0.06 to 0.31]

10. Secondary Outcome: Mean eGFR at Week 52 Based on CKD-EPI Creatinine Equation
Description: Mean eGFR at Week 52 calculated by CKD-EPI creatinine equation
Time Frame: Measured at Week 52 Post-transplant
Population: Full Analysis Population participants with available data at Week 52
Measure: Mean (95% Confidence Interval); unit: mL/min/1.73 m²
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 44 | 37
mL/min/1.73 m² | 59.2 [53.2 to 65.2] | 49.3 [43.5 to 55.1]

11. Secondary Outcome: The Slope of eGFR Over Time in Year 1
Description: The slope of eGFR over time in Year 1, calculated by CKD-EPI Creatinine equation. Slope is computed via the repeated measures analysis, covering the study time points of weeks 13, 26, 39 and 52. The estimated average slope (and corresponding 95% confidence interval) is provided for incremental progression from one time point to the next (i.e., the displayed slope shows the extent of increase (positive) or decrease (negative) in eGFR level per every time point (13 weeks) elapsed.
Time Frame: Time points in Year 1 (four time points: weeks 13, 26, 39, 52)
Population: Participants from the Full Analysis Population with available eGFR data in Year 1.
Measure: Mean (95% Confidence Interval); unit: mL/min/1.73 m² per 13 weeks
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 47 | 42
mL/min/1.73 m² per 13 weeks | -0.1 [-1.6 to 1.5] | -0.5 [-2.2 to 1.2]

12. Secondary Outcome: HIV DNA in Peripheral Blood CD4+ T Cells at Week 52
Description: HIV DNA in peripheral blood CD4+ T cells at Week 52. The standard ACTG type extraction protocol was used to extract DNA from PBMC. The readout was copies of cellular HIV-1 DNA per million PBMC. Subsequently, the outcome measure/value was obtained by multiplying the readout by the participant's CD4 percentage level at that time point, to obtain the measure of copies of HIV-1 DNA per million peripheral blood CD4+ T cells
Time Frame: At week 52 post-transplant
Population: Full Analysis Population
Measure: Median (Inter-Quartile Range); unit: copies of HIV-1 DNA/million CD4+ T cells
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 33 | 24
copies of HIV-1 DNA/million CD4+ T cells | 22.2 [4.1 to 68.4] | 43.9 [12.6 to 89.4]

13. Secondary Outcome: HIV RNA in Peripheral Blood CD4+ T Cells at Week 52.
Description: HIV RNA in peripheral blood CD4+ T cells at Week 52. The standard ACTG type extraction protocol was used to extract RNA from PBMC. The readout was copies of cellular HIV-1 RNA per million PBMC. Subsequently, the outcome measure/value was obtained by multiplying the readout by the participant's CD4 percentage level at that time point, to obtain the measure of copies of HIV-1 RNA per million peripheral blood CD4+ T cells
Time Frame: Week 52 Post Transplant
Population: Full Analysis Population
Measure: Median (Inter-Quartile Range); unit: copies of HIV-1 RNA/million CD4+ T cells
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 24 | 22
copies of HIV-1 RNA/million CD4+ T cells | 402.1 [43.5 to 2631.8] | 902.6 [191.3 to 5788.3]

14. Secondary Outcome: Plasma HIV RNA Levels (Single Copy Assay) at Week 52
Description: Plasma HIV RNA levels (single copy assay) at Week 52 Post-transplant
Time Frame: Week 52 Post-transplant
Population: Full Analysis Population
Measure: Median (Inter-Quartile Range); unit: copies of HIV-1 RNA/mL
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 29 | 28
copies of HIV-1 RNA/mL | 0 [0 to 1.3] | 0.3 [0 to 0.6]

15. Secondary Outcome: Cumulative Incidence/Proportion of Biopsy Proven Acute Rejection Within 1 Year Post Transplant
Description: Defined by histologic evidence of rejection and graft dysfunction as identified on central read of biopsy slides as well as on site biopsies. When a central read of biopsy slide is available, those results will be used; in its absence, site biopsy result will be used. Both acute cellular and humoral rejections were considered for this outcome measure, but borderline results were excluded.
Time Frame: Within Year 1 Post-transplant
Population: Full Analysis Population
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 49 | 48
Proportion of participants | 0.0816 [0.0319 to 0.2088] | 0.1250 [0.0591 to 0.2642]

16. Secondary Outcome: Cumulative Incidence/Proportion of Acute Cellular Rejection Grade Equal to or Greater Than 1A During the Entire Study Follow-up
Description: Measured by the Banff 2007 criteria as identified on central read of biopsy slides; for site biopsy results, grading was not available, all results except for borderline results were assumed to be grade 1A or greater. If available, central read result was used; if not, site biopsy result was used.
Time Frame: Within 3 years post-transplant
Population: Full Analysis Population
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 49 | 48
Proportion of participants | 0.1224 [0.0579 to 0.2591] | 0.1429 [0.0720 to 0.2836]

17. Secondary Outcome: Incidence/Proportion of Antibody Mediated Rejection
Description: Incidence of humoral/antibody mediated rejection within 52 weeks of the transplant. Both central reads and site biopsy results were included, and central read result was used if one was available, and if not, the site biopsy result was used.
Time Frame: Within 52 weeks post transplant
Population: Full Analysis Population
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 49 | 48
Proportion of participants | 0.0000 [0.0000 to NA] — Upper 95% Confidence Limit was not estimable. | 0.0208 [0.0030 to 0.1449]

18. Secondary Outcome: Proportion of Participants With de Novo Anti-donor Human Leukocyte Antigen (HLA) Antibodies
Description: Proportion of participants with de novo anti-donor human leukocyte antigen (HLA) antibodies at Week 52
Time Frame: Measured at Week 52
Population: Full Analysis Population with participants contributing data to week 52 time point
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 25 | 23
Proportion of participants | 0.1600 [0.0652 to 0.3928] | 0.0870 [0.0231 to 0.3269]

19. Secondary Outcome: Incidence/Proportion of Participants With HIV Infection in the Renal Allograft
Description: Histology/in situ hybridization was used to assess HIV infection in the renal allograft and calculate the proportion of participants with HIV infection
Time Frame: Month 6 Post-transplant
Population: Full Analysis Population
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 15 | 10
Proportion of participants | 0 [0 to NA] — Upper 95% Confidence Limit was not estimable | 0 [0 to NA] — Upper 95% Confidence Limit was not estimable

20. Secondary Outcome: Incidence of Death at Year 1
Description: Incidence of death within Year 1 post-transplant
Time Frame: Within Year 1 Post-transplant
Population: Full Analysis Population
Measure: Number (95% Confidence Interval); unit: Percent (KM estimate for incidence)
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 49 | 48
Percent (KM estimate for incidence) | 4.3 [1.1 to 16.3] | 2.2 [0.3 to 14.7]

21. Secondary Outcome: Incidence of Graft Loss in Year 1
Description: Incidence of graft loss within Year 1 post-transplant.
Time Frame: Within Year 1 Post-transplant
Population: Full Analysis Population
Measure: Number (95% Confidence Interval); unit: Percent (KM estimate for incidence)
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 49 | 48
Percent (KM estimate for incidence) | 6.3 [2.1 to 18.2] | 6.6 [2.2 to 19.0]

22. Secondary Outcome: Incidence of All Adverse Events (AEs) Greater Than or Equal to Grade 3 at Year 1
Description: Incidence of all adverse events (AEs) greater than or equal to Grade 3 within 1 year post-transplant
Time Frame: Within Year 1 Post-transplant
Population: Full Analysis Population
Measure: Number (95% Confidence Interval); unit: Percent (KM estimate for incidence)
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 49 | 48
Percent (KM estimate for incidence) | 81.6 [69.8 to 90.9] | 77.6 [64.9 to 88.2]

23. Secondary Outcome: Incidence of Serious Adverse Events (SAEs) Greater Than or Equal to Grade 3 Within Year 1
Description: Incidence of serious adverse events (SAEs) greater than or equal to Grade 3 within 1 year post-transplant
Time Frame: Within Year 1 Post-transplant
Population: Full Analysis Population
Measure: Number (95% Confidence Interval); unit: Percent (KM estimate for incidence)
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 49 | 48
Percent (KM estimate for incidence) | 73.5 [60.7 to 84.8] | 53.2 [39.8 to 68.0]

24. Secondary Outcome: Incidence of Opportunistic Infections or Neoplasms Within Year 1
Description: Incidence of opportunistic infections or neoplasms within 1 year post-transplant
Time Frame: Within Year 1 Post-transplant
Population: Full Analysis Population
Measure: Number (95% Confidence Interval); unit: Percent (KM estimate for incidence)
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 49 | 48
Percent (KM estimate for incidence) | 19.1 [10.4 to 33.5] | 6.7 [2.2 to 19.4]

25. Secondary Outcome: Incidence of Non-opportunistic Infections Requiring Hospitalization Within Year 1
Description: Incidence of non-opportunistic infections requiring hospitalization within 1 year post-transplant
Time Frame: Within Year 1 Post-transplant
Population: Full Analysis Population
Measure: Number (95% Confidence Interval); unit: Percent (KM estimate for incidence)
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 49 | 48
Percent (KM estimate for incidence) | 21.3 [12.1 to 36.1] | 28.6 [17.7 to 44.2]

26. Secondary Outcome: Calcineurin Inhibitor (Tacrolimus) Trough Levels for Participants on Maraviroc Versus Placebo
Description: Calcineurin inhibitor (tacrolimus) trough levels, from 0-12 hours post-dose at month 3 post-transplant for a subset of participants enrolled at UCSF
Time Frame: Month 3 Post-transplant (0-12 hours post-dose)
Population: PK Analysis Population: Subset of Participants Enrolled at UCSF
Measure: Median (Inter-Quartile Range); unit: nM
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 8 | 5
nM | 9.70 [8.56 to 12.30] | 12.10 [11.6 to 12.7]

27. Secondary Outcome: Calcineurin Inhibitor (Tacrolimus) AUC for Participants on Maraviroc Versus Placebo
Description: Calcineurin inhibitor (tacrolimus) AUC, 0-12 hours post-dose at month 3 post-transplant for a subset of participants enrolled at UCSF
Time Frame: Month 3 Post-transplant (0-12 hours post-dose)
Population: PK Analysis Population: Subset of participants enrolled at UCSF
Measure: Median (Inter-Quartile Range); unit: nmol-h/L
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
Number analyzed (Participants) | 8 | 5
nmol-h/L | 191.17 [160.00 to 210.14] | 193.22 [190.78 to 206.82]

28. Secondary Outcome: AUC of CCR5 Blockade (Maraviroc)
Description: AUC of CCR5 blockade (maraviroc), 0-12 hours post-dose at month 3 post-transplant in a subset of participants enrolled at UCSF
Time Frame: Month 3 Post-transplant (0-12 hours post-dose)
Population: PK Analysis Population: Maraviroc recipients in a subset of participants enrolled at UCSF
Measure: Median (Inter-Quartile Range); unit: nmol-h/L
Arm/Group | Arm 1: Maraviroc (MVC)
Number analyzed (Participants) | 8
nmol-h/L | 3101.82 [2700.76 to 5892.17]

29. Secondary Outcome: Trough Levels of CCR5 Blockade (Maraviroc)
Description: Trough levels of CCR5 blockade (maraviroc) from 0-12 hours post-dose testing at month 3 post-transplant in a subset of participants enrolled at UCSF
Time Frame: Month 3 Post-transplant (0-12 hours post-dose)
Population: PK Analysis Population: Maraviroc recipients in a subset of participants enrolled at UCSF
Measure: Median (Inter-Quartile Range); unit: nM
Arm/Group | Arm 1: Maraviroc (MVC)
Number analyzed (Participants) | 8
nM | 90.95 [73.75 to 170.00]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study follow-up period of up to ~ 3 years post-transplant. Adverse events will be collected from the time of transplant until a participant completes study participation or until 30 days after he/she prematurely withdraws (without withdrawing consent) or is withdrawn from the study.
Description: Clinicaltrials.gov definitions of AEs were followed. Only grade 3 or higher AEs were required to be recorded in the database. However, all cases of the following should be recorded, regardless of grade:
  * Postural hypotension
  * Allergic reaction
  * Rash
  * HIV persistent virologic failure defined as an HIV viral load >1000 copies/mL for more than 90 days that is not the result of an investigator/physician approved interruption in antiretroviral treatment.
Arm/Group | Arm 1: Maraviroc (MVC) | Arm 2: Placebo
All-Cause Mortality (participants affected / at risk) | 5/49 | 3/48
Serious Adverse Events (participants affected / at risk) | 37/49 | 34/48
Other Adverse Events (participants affected / at risk) | 28/49 | 37/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Maraviroc (MVC) (N=49) | Arm 2: Placebo (N=48)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0
Ileal perforation (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Retroperitoneal effusion (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 3
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Kidney transplant rejection (Immune system disorders) | 1 | 1
Transplant rejection (Immune system disorders) | 5 | 2
Abdominal abscess (Infections and infestations) | 0 | 1
Arthritis infective (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 2
COVID-19 (Infections and infestations) | 6 | 7
COVID-19 pneumonia (Infections and infestations) | 4 | 4
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 1
Gastroenteritis cryptosporidial (Infections and infestations) | 1 | 0
Gastroenteritis shigella (Infections and infestations) | 1 | 0
Mycotic endophthalmitis (Infections and infestations) | 0 | 1
Neurosyphilis (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Primary syphilis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 3 | 3
Renal graft infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Syphilis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 6
Urosepsis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 0 | 2
Delayed graft function (Injury, poisoning and procedural complications) | 1 | 2
Graft loss (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Product administration interrupted (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 3 | 0
Blood glucose increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 2 | 1
SARS-CoV-2 test positive (Investigations) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Mucoepidermoid carcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 5
Anuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Perinephric collection (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Subcapsular renal haematoma (Renal and urinary disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Diabetic bullosis (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Pancreas transplant (Surgical and medical procedures) | 0 | 1
Arteriovenous fistula (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypertensive urgency (Vascular disorders) | 1 | 0
Iliac artery dissection (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Maraviroc (MVC) (N=49) | Arm 2: Placebo (N=48)
Transplant rejection (Immune system disorders) | 5 | 2
COVID-19 pneumonia (Infections and infestations) | 4 | 3
Pyelonephritis (Infections and infestations) | 3 | 3
Urinary tract infection (Infections and infestations) | 2 | 6
Blood creatinine increased (Investigations) | 12 | 7
Blood glucose increased (Investigations) | 8 | 6
Glomerular filtration rate abnormal (Investigations) | 5 | 7
Haemoglobin decreased (Investigations) | 14 | 11
Lymphocyte count decreased (Investigations) | 3 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 7
Acute kidney injury (Renal and urinary disorders) | 3 | 5
Haematuria (Renal and urinary disorders) | 3 | 2
Hypertension (Vascular disorders) | 5 | 4

LIMITATIONS AND CAVEATS:
For the primary outcome "measured GFR by iohexol clearance at week 52", only 30 subjects (vs. 130 planned) could complete the on-site iohexol study due to COVID-19 restrictions and contribute data. There were also consistency/reliability issues with the generated data due to varying laboratory controls. Secondary outcome of "Mean eGFR at Week 52 Based on CKD-EPI Creatinine Equation" is a good surrogate for the primary outcome, with better reliability and bigger sample size for group comparison.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT02741323/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT02741323/ICF_001.pdf